CLINICAL TRIAL: NCT02110485
Title: Randomized Controlled Trial of a Patient Activation Tool in Pediatric Appendicitis to Determine Choice Between Antibiotics Alone vs. Appendectomy
Brief Title: Randomized Controlled Trial of a Patient Activation Tool in Pediatric Appendicitis (Antibiotics Alone vs. Appendectomy)
Acronym: Appy-PAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peter Minneci (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor-Investigator, Peter Minneci, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB13-00335; 4350 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2014-03-10; First posted 2014-04-10 (Estimated); Results first posted 2019-07-11 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Appendicitis; Children
Keywords: Appendicitis; Pediatric; Children; Non-operative; Antibiotics alone
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient Activation Tool (Experimental): Patients and their caregivers will receive the patient activation tool in addition to standard consultation
  Interventions: Other: Patient Activation Tool
- Standard Consultation (No Intervention): Patients and their caregivers will receive standard consultation alone

INTERVENTIONS:
Other: Patient Activation Tool — An interactive tablet based tool designed to (1) teach patient activation strategies; (2) provide evidence-based information about a health condition, (3) help patient/caregiver dyads recognize and clarify their own values, and (4) provide guidance in decision making and communication among those involved with the decision.
  Arms: Patient Activation Tool

SUMMARY:
The purpose of this study is to determine if a patient activation tool (PAT) can improve decision making and patient centered outcomes in pediatric patients with appendicitis and their caregivers choosing between antibiotics alone and appendectomy.

DETAILED DESCRIPTION:
The objective of this study is to to determine if a patient activation tool (PAT) can improve decision making and patient centered outcomes in pediatric patients with appendicitis and their caregivers.

Hypothesis: A PAT that activates patient-caregiver dyads will improve decision making and patient centered outcomes without compromising medical outcomes in children with appendicitis. Specifically,the investigators expect the PAT to improve decision self-efficacy and healthcare satisfaction without increasing disability days.

Methods/Outcomes: The investigators will perform a randomized controlled trial comparing a PAT to standard surgical consultation in patient-caregiver dyads choosing between either antibiotics alone or appendectomy for early appendicitis. The investigators will identify differences in various components of decision making and patient centered outcomes including caregiver decision self-efficacy, preparedness for decision making, decisional conflict, decision regret, caregiver activation, caregiver and child satisfaction with care and health related quality of life (HRQOL), and caregiver and child knowledge. The investigators will also characterize the effects of a PAT on medical outcomes from appendicitis in patients receiving the PAT compared to those receiving standard surgical consultation alone. The investigators will determine differences in disability days, length of stay, readmission rates, and medical complications related to treatment choice (e.g. infection, recurrence).

ELIGIBILITY:
Inclusion Criteria:

* Age : 7-17 years
* Ultrasound (US) or Computed Tomography (CT) confirmed early appendicitis:

  * US: hyperemia, <1.1 cm in diameter, compressible or non-compressible, no abscess, no fecalith, no phlegmon
  * CT: hyperemia, fat stranding, <1.1 cm in diameter, no abscess, no fecalith, no phlegmon
* White Blood Cell count < 18,000
* C-reactive Protein<4 (if obtained)
* Focal abdominal pain </= 48 hours prior to receiving antibiotics

Exclusion Criteria:

* Positive urine pregnancy test
* Other significant co-morbidities:

  * cardiovascular disease
  * malignancy
  * pulmonary disease
  * severe developmental delay

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2019-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine J Deans, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Minneci PC, Nacion KM, Lodwick DL, Cooper JN, Deans KJ. Improving Surgical Research by Involving Stakeholders. JAMA Surg. 2016 Jun 1;151(6):579-80. doi: 10.1001/jamasurg.2015.4898. No abstract available. PMID 26865380
- [Derived] Minneci PC, Cooper JN, Leonhart K, Nacion K, Sulkowski J, Porter K, Wei L, Deans KJ. Effects of a Patient Activation Tool on Decision Making Between Surgery and Nonoperative Management for Pediatric Appendicitis: A Randomized Clinical Trial. JAMA Netw Open. 2019 Jun 5;2(6):e195009. doi: 10.1001/jamanetworkopen.2019.5009. PMID 31173118

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patient Activation Tool | Standard Consultation
Started | 98 | 102
Completed | 91 | 83
Not Completed | 7 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient Activation Tool | Standard Consultation | Total
Number analyzed (Participants) | 98 | 102 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 98 | 102 | 200
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 12 [10 to 14] | 13 [9 to 15] | 12 [9 to 15]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 41 | 80
  Male | 59 | 61 | 120
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 7 | 13
  White | 88 | 85 | 173
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 0 | 5 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 98 | 102 | 200
Insurance Status [Count of Participants; unit: Participants]
  Private Insurance | 59 | 67 | 126
  Medicaid | 37 | 28 | 65
  No insurance | 2 | 7 | 9

OUTCOME MEASURES:

1. Primary Outcome: Decision Self-Efficacy Scale
Description: Decision Self-Efficacy will be measured using the Decision Self-Efficacy Scale which measures the participant's confidence in their ability to make decisions and consists of 11 questions regarding different aspects of decision making. This will be measured 1 hour after treatment decision has been made. The scale is a 5 point scale ranging from 0-not at all confident to 4-very confident. Higher scores are better.
  Scoring includes summing all items, dividing by 11; and multiplying by 25. A score of 0 means "extremely low self efficacy and a score of 100 means extremely high self efficacy
Time Frame: 1 hour following decision
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Patient Activation Tool | Standard Consultation
Number analyzed (Participants) | 98 | 102
units on a scale | 100 [95.5 to 100] | 100 [97.7 to 100]
Statistical Analysis 1: Comparison: Patient Activation Tool vs Standard Consultation; Test type: Superiority; p = 0.03, Wilcoxon (Mann-Whitney)

2. Primary Outcome: PedsQL 3.0 Healthcare Satisfaction Generic Module (Parent Report)
Description: Healthcare satisfaction will be measured at the time of discharge (average 1-2 days) using the PedsQL 3.0 Healthcare Satisfaction Generic Module- Parent Report. This survey measures the parent's satisfaction with the care their child received and measures six dimensions (information, inclusion of family, communication, technical skills, emotional needs, and overall satisfaction) using 24 items. Parents chose a score from 0-4; 0=never happy; 1=sometimes happy; 2=often happy; 3=almost always happy; 4=always happy, followed by the ability to respond "not applicable"
  Subscale scores are not reported
  If not applicable is chosen, the item is not scored nor included n the final sum. Scoring is based on a total sum for all items as well as a subscale sum for each of the 6 dimensions. Higher scores are better. Total scores range from 0-96
Time Frame: 1 day from enrollment
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Patient Activation Tool | Standard Consultation
Number analyzed (Participants) | 98 | 102
units on a scale | 98.3 [91.7 to 100] | 99.0 [94.7 to 100]
Statistical Analysis 1: Comparison: Patient Activation Tool vs Standard Consultation; Test type: Other; p = .27, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Disability Days
Description: Disability days will be assessed at 1 year follow-up. Disability days is a composite of inpatient hospital days, emergency department visits, primary care physician visits and all days with limited activities referable to their appendicitis.
Time Frame: 1 year folow-up
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Patient Activation Tool | Standard Consultation
Number analyzed (Participants) | 83 | 91
Days | 5 [2 to 15] | 6 [2 to 11]
Statistical Analysis 1: Comparison: Patient Activation Tool vs Standard Consultation; Test type: Other; p = .67, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Patient Activation Measure (PAM)
Description: Parent activation will be assessed with the Patient Activation Measure® (Parent-PAM®) using a version of healthy child parent PAM® adapted with permission. This 13 item scale and was derived from the short form version of the Patient Activation Measure®. The Parent-PAM® is used to assess the parent's activation in the management of their child's health.
  The 13 items have response options ranging from 1=strongly disagree to 4 strongly agree with an option to respond as "not applicable". A total PAM score is calculated by summing all items and dividing by the number of items answered and multiplied by 13; total scores can range from 13-52. This score is transformed to a scale ranging from 0-100 with higher PAM scores indicating higher patient activation.
Time Frame: 1 hour
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Patient Activation Tool | Standard Consultation
Number analyzed (Participants) | 98 | 102
units on a scale | 91 [75 to 100] | 100 [77.7 to 100]
Statistical Analysis 1: Comparison: Patient Activation Tool vs Standard Consultation; Test type: Other; p = .17, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Number of Participants Readmitted
Description: Readmissions rates to any hospital within 1 year wil be assessed
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Activation Tool | Standard Consultation
Number analyzed (Participants) | 83 | 91
Participants | 15 | 15
Statistical Analysis 1: Comparison: Patient Activation Tool vs Standard Consultation; Test type: Other; p = .84, Fisher Exact

6. Secondary Outcome: PedsQL Pediatric Quality of Life Inventory and PedsQL Family Impact Module Scales
Description: The PedsQL Pediatric Quality of Life Inventory is a 23 item survey with response options offered on a 5 point scale; 0= never been a problem; 1=almost never a problem; 2=sometimes a problem; 3=often a problem; 4=almost always a problem. A total score is summed for each of the 4 dimensions as well as an overall score for the entire measure.
  The PedsQL Family Impact Module Scales include subscales: physical functioning; emotional functioning; social functioning; cognitive functioning; communication; worry; family functioning; daily activities; and family relationships. The options for this 5-point scale range from 0= never a problem to 4=always a problem). Items are reverse-scored and high scores indicate better family functioning. A total summed score is utilized. Each subscale can be summed individually and divided by the number of items in that.
  Total scores for this measure range from 0-92
Time Frame: 30 day follow-up
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Patient Activation Tool | Standard Consultation
Number analyzed (Participants) | 71 | 76
units on a scale | 88.0 [79.3 to 96.7] | 88.0 [81.0 to 96.7]
Statistical Analysis 1: Comparison: Patient Activation Tool vs Standard Consultation; Test type: Other; p = .99, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration of the study. Adverse events per participant were tracked up through the completion of their last time point, 1 year post-enrollment.
Arm/Group | Patient Activation Tool | Standard Consultation
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/102
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/102
Other Adverse Events (participants affected / at risk) | 0/98 | 0/102

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2017-02-06): https://cdn.clinicaltrials.gov/large-docs/85/NCT02110485/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-06): https://cdn.clinicaltrials.gov/large-docs/85/NCT02110485/SAP_001.pdf
  • Informed Consent Form (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/85/NCT02110485/ICF_002.pdf